CLINICAL TRIAL: NCT06859840
Title: Clinical Research on the Use of Abdominal CT Combined With AI for Early Screening
Brief Title: Abdominal CT Combined With AI for Early Screening of Liver Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: LIDAR
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Artificial Intelligence; Hepatocellular Carcinoma; LIDAR
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: The AI model will be used to identify imaging findings suggestive of liver space-occupying lesions. Senior liver specialists from our hospital's hepatobiliary-pancreatic surgery and radiology departments, who have expertise in AI research and clinical application, will delineate these liver lesions in conjunction with pathological results to develop and refine the model. After model establishment, external multicenter validation will be conducted to assess the model's stability in detecting focal liver lesions across diverse populations. For cases where the model indicates malignancy without clear evidence from medical history or other data, follow-up will be performed to confirm the true value through pathological results. The primary focus will be to evaluate whether the model can improve the detection rate of focal liver lesions requiring intervention in various complex real-world scenarios.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIDAR (Experimental)
  Interventions: Device: LIDAR
- Control (No Intervention)

INTERVENTIONS:
Device: LIDAR — Using the LIDAR model to assist in image interpretation, patients with positive results are recalled for further examination based on the LIDAR output information and the original image interpretation, to obtain pathological results and long-term follow-up.
  Arms: LIDAR

SUMMARY:
This study plans to utilize multiphase contrast-enhanced and non-contrast CT（Computed Tomography） images from 10000 pathologically confirmed liver tumor patients at our hospital. An AI（artificial intelligence） model will be used to outline the 3D contours of liver masses, which will then be refined by radiologists and hepatobiliary-pancreatic surgeons to enhance model accuracy. By incorporating more imaging data, the model's recognition capabilities will be improved, laying the groundwork for prospective clinical trials and aiming to establish a superior AI model for early liver cancer screening based on CT imaging.

DETAILED DESCRIPTION:
This research project intends to utilize multiphase contrast-enhanced and non-contrast CT images from 10000 patients with a full spectrum of liver tumors (such as HCC（hepatocellular carcinoma）, ICC（intrahepatic cholangiocarcinoma ）, META（Metastasis）, etc.), confirmed by the pathological gold standard at our hospital. Through a pre-established AI model, the 3D contours of various liver masses will be delineated. In collaboration with senior physicians from our hospital's radiology department and hepatobiliary pancreatic surgery department, the AI-drawn contours will be refined to obtain more accurate 3D mass models, thereby enhancing the validation efficacy of the model. By incorporating more radiological data, the precision of the model will be improved, boosting its recognition capabilities and laying a solid foundation for subsequent prospective clinical trials. The ultimate goal is to establish a superior AI model for early screening of liver cancer based on CTimaging.

ELIGIBILITY:
Inclusion Criteria:

* From 2019 to 2030, our hospital has collected non-contrast and contrast-enhanced CT images from patients with a full spectrum of liver tumors (such as HCC, ICC, META, etc.), all confirmed by the pathological gold standard

Exclusion Criteria:

* Patients who have undergone upper abdominal surgery. Examples include post-ERCP (Endoscopic Retrograde Cholangiopancreatography) for the pancreas, post-external drainage surgery, esophageal surgery, and gastrectomy, among others.
* Patients who have received systemic treatments such as chemotherapy or traditional Chinese medicine. Examples include chemotherapy for lymphoma, chemotherapy for leukemia, chemotherapy for lung cancer, and comprehensive treatment for liver cancer, etc.
* Patients with poor-quality CT images. Examples include convolution artifacts caused by the inability to place hands on the sides of the body and respiratory artifacts due to poor breath-holding, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2030-03-15 (Estimated); Study Completion 2030-09-15 (Estimated)

PRIMARY OUTCOMES:
Detection efficiency in liver tumor assisted by LIDAR | Complete the statistics within six months after the patient is fully enrolled, and it is expected to take 2 years from the start of the study
  Sensitivity、Specificity
Detection efficiency in liver tumor assisted by LIDAR | Complete the statistics within six months after the patient is fully enrolled, and it is expected to take 2 years from the start of the study
  PPV、NPV
Detection efficiency in liver tumor assisted by LIDAR | Complete the statistics within six months after the patient is fully enrolled, and it is expected to take 2 years from the start of the study
  AUC

SECONDARY OUTCOMES:
TNM stage | 1 day (evaluate through CT imaging before surgery)
  Staging of liver cancer
OS | From diagnosis of liver cancer to 5 years later
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No